CLINICAL TRIAL: NCT07315594
Title: Cluster Randomized Trial of Initial Oxygen Concentration at Birth in Late-Preterm Infants
Brief Title: Initial Oxygen Concentration at Birth in Late-Preterm Infants
Acronym: OXY-PREEM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro00146615
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth | interventions — Oxygen

STUDY DESIGN:
Intervention Model Description: This will be a cluster-crossover design, unmasked randomized controlled trial (RCT) comparing two oxygen concentrations at initiation of resuscitation.
Masking Description: Blinding will not be feasible, as each center will be assigned to each study intervention and then switch to the second intervention group. However, the trial statistician and DSMB will be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Initial use of 60% oxygen during breathing support in the delivery room (Experimental): Infants randomized to the 60% Oxygen (FiO₂) Group will begin respiratory support with an initial inspired oxygen concentration of 60%. At birth, all infants will receive 60 seconds of delayed cord clamping as standard care. Following cord clamping, a pulse oximeter will be applied to measure peripheral oxygen saturation (SpO₂), with a reliable signal typically available at approximately 3 minutes of age.
  At 3 minutes of age, the clinical team will assess SpO₂. If SpO₂ is <85%, the inspired oxygen concentration will be increased by 20% every 60 seconds to achieve an SpO₂ >85% by 5 minutes of age. If SpO₂ is >95% at or before 5 minutes of age, the inspired oxygen concentration will be decreased stepwise in increments of 10-20% every 60 seconds to maintain an SpO₂ >85% between 5 and 10 minutes of age, or an SpO₂ of 90-95% at and beyond 10 minutes of age.
  Interventions: Drug: 60% Oxygen Group - Infants will start in 60% oxygen
- Initial use of 30% oxygen during breathing support in the delivery room (Active Comparator): Infants randomized to the 30% Oxygen (FiO₂) Group will begin respiratory support with an initial inspired oxygen concentration of 30%. At birth, all infants will receive 60 seconds of delayed cord clamping as standard care. Following cord clamping, a pulse oximeter will be applied to measure peripheral oxygen saturation (SpO₂), with a reliable signal typically available at approximately 3 minutes of age.
  At 3 minutes of age, the clinical team will assess SpO₂. If SpO₂ is <85%, the inspired oxygen concentration will be increased by 20% every 60 seconds to achieve an SpO₂ >85% by 5 minutes of age. If SpO₂ is >95% at or before 5 minutes of age, the inspired oxygen concentration will be decreased stepwise in increments of 10-20% every 60 seconds to maintain an SpO₂ >85% between 5 and 10 minutes of age, or an SpO₂ of 90-95% at and beyond 10 minutes of age.
  Interventions: Drug: 30% Oxygen Group - Infants will start in 30% oxygen

INTERVENTIONS:
Drug: 60% Oxygen Group - Infants will start in 60% oxygen — Infants randomized to the 60% Oxygen (FiO₂) Group will begin respiratory support with an initial inspired oxygen concentration of 60%. At birth, all infants will receive 60 seconds of delayed cord clamping as standard care. Following cord clamping, a pulse oximeter will be applied to measure peripheral oxygen saturation (SpO₂), with a reliable signal typically available at approximately 3 minutes of age.
  At 3 minutes of age, the clinical team will assess SpO₂. If SpO₂ is <85%, the inspired oxygen concentration will be increased by 20% every 60 seconds to achieve an SpO₂ >85% by 5 minutes of age. If SpO₂ is >95% at or before 5 minutes of age, the inspired oxygen concentration will be decreased stepwise in increments of 10-20% every 60 seconds to maintain an SpO₂ >85% between 5 and 10 minutes of age, or an SpO₂ of 90-95% at and beyond 10 minutes of age.
  Other Names: 60% Oxygen Group
  Arms: Initial use of 60% oxygen during breathing support in the delivery room
Drug: 30% Oxygen Group - Infants will start in 30% oxygen — Infants randomized to the 30% Oxygen (FiO₂) Group will begin respiratory support with an initial inspired oxygen concentration of 30%. At birth, all infants will receive 60 seconds of delayed cord clamping as standard care. Following cord clamping, a pulse oximeter will be applied to measure peripheral oxygen saturation (SpO₂), with a reliable signal typically available at approximately 3 minutes of age.
  At 3 minutes of age, the clinical team will assess SpO₂. If SpO₂ is <85%, the inspired oxygen concentration will be increased by 20% every 60 seconds to achieve an SpO₂ >85% by 5 minutes of age. If SpO₂ is >95% at or before 5 minutes of age, the inspired oxygen concentration will be decreased stepwise in increments of 10-20% every 60 seconds to maintain an SpO₂ >85% between 5 and 10 minutes of age, or an SpO₂ of 90-95% at and beyond 10 minutes of age.
  Other Names: 30% Oxygen Group
  Arms: Initial use of 30% oxygen during breathing support in the delivery room

SUMMARY:
This study is aims to examine the best amount of oxygen to give preterm babies (born between 32 and 35 weeks) right after birth.

In the past, doctors used high levels of oxygen, but research has shown that using lower levels might help reduce the risk of death in full-term babies without harming brain development. However, investigators don't know the best oxygen level for babies born a little early (32 to 35 weeks). Some early data suggests that giving lower oxygen levels (FiO2 0.3) may not help babies reach healthy oxygen levels by 5 minutes after birth. This study will compare two oxygen levels-FiO2 0.6 and FiO2 0.3 to see which helps babies breathe better and need less ongoing breathing support. Researchers will study over 1,500 babies in hospitals across Alberta, Canada, to find the safest approach for these babies.

ELIGIBILITY:
Inclusion Criteria:

* i) Infants with gestational age between 32+0-35+6 weeks based on best available obstetrical estimate, requiring respiratory support
* ii) Infants designated to receive full resuscitation, i.e., no parental request or pre-determined decision to provide only comfort care at birth
* iii) No known major congenital or chromosomal malformation.

Exclusion Criteria:

* i) Infant born outside of study centers and transported to centers after delivery.

Ages: 0 Minutes to 10 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1520 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Need for ongoing respiratory support within the 1st hour after birth | first 60 minutes after birth
  Ongoing respiratory support will be defined as: the need for intubation and mechanical ventilation or the use of any non-invasive respiratory supports (e.g., CPAP, nasal high flow therapy or low flow oxygen) after initial resuscitation

SECONDARY OUTCOMES:
Mortality in the delivery room | first 60 minutes after birth
  Preterm infants who do not survive the resuscitation at birth
Mortality prior discharge | up to 100 days after birth
  Preterm infants who do not survive during the admission to the neonatal intensive care unit
Duration of hospital stay | up to 100 days
  duration in days the preterm infant will be admitted to the neonatal intensive care unit
Air leak | first 72 hours after birth
  Air leak defined as pneumothorax

CONTACTS AND LOCATIONS:
Overall Officials: Georg Schmolzer, Principal Investigator — University of Alberta
Locations (1):
- Royal Alexandra Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
there is no current plan, however requests can be send to Prof. Georg Schmolzer via schmolze@ualberta.ca.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The Study Protocol and the Statistical Analysis Plan (SAP) will be published during the recruitment phase of the trial.
  Informed Consent Form (ICF) and Clinical Study Report (CSR) can be requested from Prof. Georg Schmolzer via schmolze@ualberta.ca
Access Criteria: Requests can be send to Prof. Georg Schmolzer via schmolze@ualberta.ca